CLINICAL TRIAL: NCT01961544
Title: Phase IV Clinical Trial to Evaluate Safety of Eribulin in Patients With Locally Advanced or Metastatic Breast Cancer
Brief Title: Eribulin Mesylate Phase IV Clinical Trial in Korean Patients With Metastatic or Locally Advanced Breast Cancer
Acronym: ESKIMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKI-CT-1301
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Breast Neoplasms; Breast Cancer
Keywords: Breast Cancer; Metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — eribulin

ARMS (1):
- Eribulin mesylate (Experimental): 1.4 mg/m2 (as eribulin 1.23 mg/m2) day by 2-5 minutes IV on Day 1 and 8 every 21 days
  Interventions: Drug: Eribulin mesylate

INTERVENTIONS:
Drug: Eribulin mesylate — 1.4 mg/m2 (as eribulin 1.23 mg/m2) day by 2-5 minutes IV on Day 1 and 8 every 21 days

SUMMARY:
This clinical study is designed as an open, single group, multi-center, phase 4 clinical study to assess the safety of eribulin which is approved for the treatment of the patients in Korea with locally advanced or metastatic breast cancer who had received two to five prior chemotherapy regimens including anthracyclines and taxanes for advanced disease.

Subjects who meet the inclusion/exclusion criteria are administered of 1.4 mg/m2 of the investigational product intravenously in 2-5 min on day 1 and day 8 of every 21-day cycle. In case of the progression of disease, unacceptable toxicity, withdrawal of the consent, or judgment by investigator that the treatment needs to be stopped, the treatment of investigational product is stopped, and treatment termination assessment is performed within 30 days from the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female, Age greater or equal to 20 years
2. Patients with histologically or cytologically confirmed carcinoma of the breast
3. Patients with locally advance or metastatic carcinoma of the breast
4. Patients who have received two to five prior chemotherapeutic regimens including an antracycline and a taxane and 2 or more regimens for locally recurrent and/or metastatic disease
5. Patients must have proved refractory to the most recent chemotherapy on or within six (6) months of therapy
6. Patients who have assessable lesion according to RECIST v 1.1
7. Adequately maintained bone marrow function

   * absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9 /L
   * hemoglobin greater than or equal to 10.0 g/dl (a hemoglobin less than 10.0 g/dL is acceptable if it is corrected by erythropoietin or transfusion)
   * Platelet count greater than or equal to 100 x 10^9 /L
8. Adequately maintained liver function

   * Total bilirubin: less than or equal to 1.5 times the upper limits of normal (ULN) and
   * Alkaline phosphatase(ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 x ULN (in the case of liver metastases less than or equal to 5 x ULN)
9. Adequately maintained renal function

   * Serum creatinine less than or equal to 2.0 mg/dl or
   * Calculated creatinine clearance greater than or equal to 40 ml/min (Cockcroft and Gault formula)
10. Resolution of all chemotherapy or radiation-related toxicities to Grade 1 severity or lower, except for

    * alopecia
    * stable sensory neuropathy less than or equal to Grade 2
11. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
12. Life expectancy of greater than or equal to 3 months
13. Patients willing and able to comply with the study protocol for the duration of the study
14. Patients who have provided written consent to participate in this study

Exclusion Criteria

1. Patients who have received a chemotherapy, radiation, biologics, immunotherapy or hormonal therapy within three weeks before treatment start (but, palliative radiation can be enrolled)
2. Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen
3. Patients with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least four weeks before starting treatment in this study. Any signs and/or symptoms of brain metastases must be stable for at least four weeks before starting study treatment
4. Patients with meningeal carcinomatosis
5. Significant cardiovascular impairment

   * Myocardial infarction within the past six months, unstable angina, history of congestive heart failure NYHA class III or IV, or serious cardiac arrhythmia
   * QTc prolongation (Bazett's Formula greater than 480 msec) or congenital long QT syndrome
6. Severe/uncontrolled intercurrent illness/infection required administration of antibiotic injection
7. Patients who have processed a major surgery within four weeks before participation in this clinical trial
8. Patients who have had a prior malignancy within the past five years other than breast cancer (but, treated non-melanoma skin cancer and carcinoma in situ of the cervix will not be excluded)
9. Patients with known positive HIV status
10. Patients who have received genetic therapy or other investigational drug within 4 weeks before treatment start or expected to receive prohibited medication
11. Patients with prior allergies to Halichondrin B, its derivatives, active ingredient, or other diluting agent
12. Patients who have received this investigational product before registration for this study
13. Patients who are pregnant, who may possibly be pregnant, or are lactating
14. Patients who do not agree to practice contraception for the study periods
15. Patients who have participated in other clinical trial within 4 weeks before screening
16. Patients otherwise judged by investigator or sub investigator to be unsuitable for inclusion

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- South Korea (14):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan

RESULTS

PARTICIPANT FLOW:
Groups:
- Eribulin Mesylate 1.4 mg/m^2: Participants received 1.4 milligrams per meters squared (mg/m^2) eribulin mesylate intravenously over the course of 2 to 5 minutes on Day 1 and Day 8 of each 21-day cycle.
Period: Overall Study
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Started | 101
Completed | 88
Not Completed | 13
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 7
Not completed — Adverse Event | 1
Not completed — Physician Decision | 2
Not completed — Poor Tolerance | 1
Not completed — Aggravation of Steral Pain | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Number analyzed (Participants) | 101
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 50.36 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE) and Any Treatment-emergent Serious Adverse Event (SAE)
Description: An AE is defined as any harmful, untoward sign (including abnormal laboratory value, etc.), symptom, or disease in a participant administered investigational product that does not necessarily have a causal relationship with treatment. An SAE is defined as an AE that is life threatening or results in death, results in hospitalization (initial or prolonged), results in a disability (significant, persistent, or permanent change, impairment, damage or disruption in the participant's body function/structure, physical activities, or quality of life), results in a congenital anomaly, or requires intervention to prevent permanent impairment or damage. TEAEs are defined as those events that started on or after the date and time of administration of the first dose of study drug and those events that were present prior to the administration of the first dose of study drug and increased in severity during the study.
Time Frame: mean of 3.76 months
Population: Safety Set: all participants who are administered investigational product at least once for the analysis
Measure: Number; unit: Participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Number analyzed (Participants) | 101
Participants
  TEAE | 101
  Treatment-emergent SAE | 20

2. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the number of participants with complete response (CR), partial response (PR), and stable disease (SD). The Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 was used to assess the tumor response. Tumor response was evaluated by investigators. CR is defined as the disappearance of all extranodal target lesions. All pathological lymph nodes must have decreased to <10 millimeters (mm) in the short axis. PR is defined as at least a 30% decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline sum diameters. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (SLD increased by at least 20% from the smallest value on study [including baseline, if that is the smallest]. The SLD must also demonstrate an absolute increase of at least 5 mm. [Two lesions increasing from 2 mm to 3 mm, for example, does not qualify]).
Time Frame: mean of 3.76 months
Population: Full Analysis Set: participants who were administered investigational product at least once after enrollment and had at least one primary efficacy data value since Baseline
Measure: Number; unit: Participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Number analyzed (Participants) | 96
Participants
  CR | 1
  PR | 15
  SD | 33

ADVERSE EVENTS:
Groups:
- Eribulin Mesylate 1.4 mg/m^2: Participants received 1.4 milligrams per meters squared (mg/m^2) eribulin mesylate intravenously over the course of 2-5 minutes on Day 1 and Day 8 of each 21-day cycle.
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Serious Adverse Events (participants affected / at risk) | 20/101
Other Adverse Events (participants affected / at risk) | 101/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate 1.4 mg/m^2 (N=101)
Consciousness fluctuating (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Wound secretion (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate 1.4 mg/m^2 (N=101)
Neutropenia (Blood and lymphatic system disorders) | 92
Anaemia (Blood and lymphatic system disorders) | 12
Leukopenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 27
Pyrexia (General disorders) | 17
Chest pain (General disorders) | 10
Asthenia (General disorders) | 8
Mucosal inflammation (General disorders) | 8
Pain (General disorders) | 7
Chills (General disorders) | 5
Influenza like illness (General disorders) | 4
Oedema peripheral (General disorders) | 2
Peripheral swelling (General disorders) | 2
Application site pain (General disorders) | 1
Face oedema (General disorders) | 1
Localised oedema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema (General disorders) | 1
Nausea (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 9
Stomatitis (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 5
Toothache (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 46
Rash (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 16
Headache (Nervous system disorders) | 12
Neuropathy peripheral (Nervous system disorders) | 11
Dizziness (Nervous system disorders) | 7
Lethargy (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 41
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 25
Back pain (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Nasopharyngitis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 3
Cystitis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Device related infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pyuria (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 2
Eating disorder symptom (Psychiatric disorders) | 1
Aspartate aminotransferase increased (Investigations) | 8
Alanine aminotransferase increased (Investigations) | 5
Electrocardiogram QT prolonged (Investigations) | 2
Haemoglobin decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Neutrophil count increased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Pelvic pain (Reproductive system and breast disorders) | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 3
Breast pain (Reproductive system and breast disorders) | 2
Eye pain (Eye disorders) | 4
Blepharitis (Eye disorders) | 1
Dry age-related macular degeneration (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Xerophthalmia (Eye disorders) | 1
Lymphoedema (Vascular disorders) | 2
Embolism (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Oliguria (Renal and urinary disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
External ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Palpitations (Cardiac disorders) | 1
Eye injury (Injury, poisoning and procedural complications) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other